CLINICAL TRIAL: NCT01020058
Title: Randomized Controlled Trial Comparing Open Mesh Repair in Local Anesthesia to Cost-Optimized Laparoscopic Repair for Primary Inguinal Hernia
Brief Title: Randomized Study of Open Mesh Repair in Local Anesthesia Versus Cost-optimized Laparoscopic Repair for Inguinal Hernia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University Hospital (Other)
Collaborators: Uppsala County Council, Sweden (Other Government)
Responsible Party: Principal Investigator, Ursula Dahlstrand, MD, PhD, Uppsala University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004:M-360
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Hernia, Inguinal
MeSH Terms: conditions — Hernia, Inguinal | interventions — tetraethylpyrazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lichtenstein in local anesthesia (LLA) (Active Comparator): Patient operated in local anesthesia, with an anterior mesh repair according to Lichtenstein
  Interventions: Procedure: Mesh repair for primary inguinal hernia
- TEP (Active Comparator): Patient receives a totally extraperitoneal laparoscopic repair
  Interventions: Procedure: Mesh repair for primary inguinal hernia

INTERVENTIONS:
Procedure: Mesh repair for primary inguinal hernia — Open Lichtenstein repair in local anesthesia using a polypropylene mesh compared to totally extra-peritoneal laparoscopic repair using a polypropylene mesh
  Other Names: Lichtenstein (LLA); TEP

SUMMARY:
The purpose of this study is to compare the frequency of long-term post operative pain after an open mesh repair ad modum Lichtenstein performed in local anaesthesia to that after an totally extraperitoneal laparoscopic repair (TEP) for primary inguinal hernia. The investigators will also be assessing the cost for the procedures and hospital care as well as the cost for sick-leave depending on procedure performed. The study hypothesis is that the laparoscopic approach will be associated with less long term post operative pain.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral inguinal hernia
* suitable for open mesh repair in local anesthesia as well as laparoscopic repair
* ASA score I-III
* informed consent

Exclusion Criteria:

* ASA score IV (not suitable for TEP)
* bilateral hernias (laparoscopic repair preferable)
* recurrent hernia (primary repair affects preferable treatment)
* large scrotal hernias (not suitable for local anesthesia)
* earlier open lower abdominal surgery, aside from appendectomy (scarring may be a hindrance for TEP)

Ages: 20 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2006-04; Primary Completion 2012-03 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
long-term post operative pain | 6 wks, 1 year

SECONDARY OUTCOMES:
cost-effectiveness of the separate procedures | 6wks, 1year

CONTACTS AND LOCATIONS:
Overall Officials: Staffan Wollert, MD, PhD, Study Director — Uppsala University Hospital
Locations (2):
- Sweden (2):
  - Enköping Hospital, Enköping
  - Uppsala University Hospital, Uppsala

REFERENCES:
- [Derived] Westin L, Wollert S, Ljungdahl M, Sandblom G, Gunnarsson U, Dahlstrand U. Less Pain 1 Year After Total Extra-peritoneal Repair Compared With Lichtenstein Using Local Anesthesia: Data From a Randomized Controlled Clinical Trial. Ann Surg. 2016 Feb;263(2):240-3. doi: 10.1097/SLA.0000000000001289. PMID 26079901
- [Derived] Dahlstrand U, Sandblom G, Ljungdahl M, Wollert S, Gunnarsson U. TEP under general anesthesia is superior to Lichtenstein under local anesthesia in terms of pain 6 weeks after surgery: results from a randomized clinical trial. Surg Endosc. 2013 Oct;27(10):3632-8. doi: 10.1007/s00464-013-2936-1. Epub 2013 Apr 10. PMID 23572220